CLINICAL TRIAL: NCT02664337
Title: Conjoint Analysis of Patient Preferences in Joint Interventions
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00067150
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Arthritis; Femoroacetabular Impingement; Osteochondritis Dissecans; Hip Fractures; Ankle Fractures; Tibial Fractures
MeSH Terms: conditions — Arthritis; Femoracetabular Impingement; Osteochondritis Dissecans; Hip Fractures; Ankle Fractures; Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision tool (Experimental): A "decision tool" will be provided to participants who currently or previously have had one of the following 12 musculoskeletal conditions: hip arthritis, knee arthritis, ankle arthritis, hip labral tears and femoroacetabular impingement (FAI), osteochondritis dissecans, Achilles tendon rupture, patellofemoral dislocation, distal radius fracture, and fractures of the hip, ankle, tibia, and proximal humerus.
  Interventions: Other: Decision tool
- Standard treatment information (Active Comparator): "Standard treatment information" will be provided to participants who currently or previously have had one of the following 12 musculoskeletal conditions: hip arthritis, knee arthritis, ankle arthritis, hip labral tears and femoroacetabular impingement (FAI), osteochondritis dissecans, Achilles tendon rupture, patellofemoral dislocation, distal radius fracture, and fractures of the hip, ankle, tibia, and proximal humerus.
  Interventions: Other: Standard treatment information

INTERVENTIONS:
Other: Decision tool — A survey will be created for each condition that reflects the most important aspects of the corresponding treatment process.
  Arms: Decision tool
Other: Standard treatment information — Participants will receive information pertaining to one of the 12 specified musculoskeletal conditions. This information will reflect information commonly distributed to patients seeking to make a decision concerning treatment for their condition.
  Arms: Standard treatment information

SUMMARY:
This study is an observational study to test and validate a questionnaire and statistical model used to determine patient preferences regarding treatment for any one of 11 musculoskeletal conditions: hip arthritis, knee arthritis, hip labral tears and femoroacetabular impingement (FAI), osteochondritis dissecans, Achilles tendon rupture, patellofemoral dislocation, distal radius fracture, and fractures of the hip, ankle, tibia, and proximal humerus. This study aims to understand how multiple treatment variables, including pain, rehabilitation time, cost, and choice of surgical versus non-surgical intervention, impact patients' decision-making processes and ultimate choice of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient age criteria for each condition is listed below:

  1. Hip arthritis: 50-80 years
  2. Knee arthritis: 50-80 years
  3. Hip labral tears and FAI: 18-65
  4. Osteochondritis dissecans: parents with children between the ages of 8-18
  5. Achilles tendon rupture: 25-60 years
  6. Patellofemoral dislocation: parents with children between the ages of 8-18 and adults between 18-50 years of age
  7. Distal radius fracture: 18-80 years
  8. Hip fracture: 50-85 years
  9. Ankle fracture: 18-80 years
  10. Tibia fracture: 18-80 years
  11. Proximal humerus fracture: 18-80 years
  12. Ankle Arthritis: 40-80 years

      Exclusion Criteria:
* Inability to read, understand and give effective English consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2310 (Estimated)
Dates: Start 2016-02; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Patient preferences survey - Hip Arthritis | 3-5 years
  Patient-voiced preferences regarding treatment for hip arthritis based on questionnaires
Patient preferences survey - Knee Arthritis | 2 years
  Patient-voiced preferences regarding treatment for knee arthritis based on questionnaires
Patient preferences survey - hip labral tears and FAI | 3-5 years
  Patient-voiced preferences regarding treatment for hip labral tears and femoroacetabular impingement (FAI) based on questionnaires
Patient preferences survey - Osteochondritis dissecans | 3-5 years
  Patient-voiced preferences regarding treatment for osteochondritis dissecans based on questionnaires
Patient preferences survey - Achilles tendon rupture | 2 years
  Patient-voiced preferences regarding treatment for Achilles tendon rupture based on questionnaires
Patient preferences survey - patellofemoral dislocation | 2 years
  Patient-voiced preferences regarding treatment for patellofemoral dislocation based on questionnaires
Patient preferences survey - distal radius fracture | 3-5 years
  Patient-voiced preferences regarding treatment for distal radius fracture based on questionnaires
Patient preferences survey - hip fracture | 3-5 years
  Patient-voiced preferences regarding treatment for hip fracture based on questionnaires
Patient preferences survey - ankle fracture | 3-5 years
  Patient-voiced preferences regarding treatment for ankle fracture based on questionnaires
Patient preferences survey - tibia fracture | 3-5 years
  Patient-voiced preferences regarding treatment for tibia fracture based on questionnaires
Patient preferences survey - proximal humerus fracture | 3-5 years
  Patient-voiced preferences regarding treatment for proximal humerus fracture based on questionnaires
Patient preferences survey - Ankle Arthritis | 3-5 years
  Patient-voiced preferences regarding treatment for ankle arthritis based on questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Mather III, MD, MBA, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No